CLINICAL TRIAL: NCT03749343
Title: International T1 Multicenter Outcome Study (the German Chapter)
Brief Title: International T1 Multicenter Outcome Study
Acronym: T1Outcome-DE
Status: Active, not recruiting | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Kerckhoff Klinik (Other)
Responsible Party: Principal Investigator, Valentina Puentmann, Principal Investigator, Clinical professor, Johann Wolfgang Goethe University Hospital
Other Study IDs: T1 Outcome 1/16gA
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Cardiomyopathies; Inflammatory Disease; Coronary Artery Disease; Chronic Kidney Diseases
Keywords: T1 mapping; native T1; native T2; accuracy; prognosis
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Coronary Artery Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mapping of magnetic relaxation within the myocardial tissue using T1 (and T2) mapping using cardiovascular magnetic resonance (CMR) are novel measures of quantifiable (scalable) myocardial tissue characterisation. Evidence suggests that myocardial mapping could be useful in detection of diffuse myocardial disease, complementing late gadolinium enhancement (LGE) as the tool for regional myocardial disease. A handful of studies, three single centre study of a single T1 index with outcomes and one multicentre study for all indices reported strong associations with all cause mortality and heart failure. These studies were based on a single-vendor platform and were using a single sequence. The main unknowns pertaining the successful translation of this technique and the transferability of the methodology beyond a single centre and lack of outcome evidence from broad and large populations. In this study, we will assess the diagnostic accuracy of T1 (and T2) mapping measurements in health and disease, and the prognostic relevance of T1 mapping measurements by associations with outcome. This study is builds upon/integrates the evidence of the NCT02407197 study, which remains active for follow-up, but is currently no longer recruiting.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>18 years of age)
2. Able to provide informed consent
3. Clinically indicated cardiac magnetic resonance imaging study

Exclusion Criteria: contraindications for clinical cardiac magnetic resonance imaging due to MR unsafe devices or objects

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults referred to clinical cardiac magnetic resonance imaging
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 year
  number of deaths
Survival | 5 year
  number of deaths

SECONDARY OUTCOMES:
Rate of Heart Failure events | 1 year
  Number of participants with events including death and Hospitalisation due to Heart Failure
Rate of Heart Failure events | 5 year
  Number of participants with events including death and Hospitalisation due to Heart Failure
Rate of Arrhythmia | 1 year
  Number of participants with events of documented Sudden Cardiac Death, appropriate ICD discharge, sustained VT
Rate of Arrhythmia | 5 year
  Number of participants with events including documented Sudden Cardiac Death, appropriate ICD discharge, sustained VT
Rate of death due to to cardiovascular causes | 1 year
  Number of participants with death due to myocardial infarction, heart failure, arrhythmia
Rate of death due to to cardiovascular causes | 5 year
  Number of participants with death due to myocardial infarction, heart failure, arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Puentmann, MD, PhD, Principal Investigator — Goethe University
Locations (2):
- Germany (2):
  - Kerckhoff Hospital, Bad Nauheim, Hesse
  - Institute for experimental and translational cardiovascular imaging, Frankfurt am Main, Hesse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Puntmann VO, Carr-White G, Jabbour A, Yu CY, Gebker R, Kelle S, Rolf A, Zitzmann S, Peker E, D'Angelo T, Pathan F, Elen, Valbuena S, Hinojar R, Arendt C, Narula J, Herrmann E, Zeiher AM, Nagel E; International T1 Multicentre CMR Outcome Study. Native T1 and ECV of Noninfarcted Myocardium and Outcome in Patients With Coronary Artery Disease. J Am Coll Cardiol. 2018 Feb 20;71(7):766-778. doi: 10.1016/j.jacc.2017.12.020. PMID 29447739
- [Result] Winau L, Hinojar Baydes R, Braner A, Drott U, Burkhardt H, Sangle S, D'Cruz DP, Carr-White G, Marber M, Schnoes K, Arendt C, Klingel K, Vogl TJ, Zeiher AM, Nagel E, Puntmann VO. High-sensitive troponin is associated with subclinical imaging biosignature of inflammatory cardiovascular involvement in systemic lupus erythematosus. Ann Rheum Dis. 2018 Nov;77(11):1590-1598. doi: 10.1136/annrheumdis-2018-213661. Epub 2018 Aug 4. PMID 30077990
- [Result] Haslbauer JD, Lindner S, Valbuena-Lopez S, Zainal H, Zhou H, D'Angelo T, Pathan F, Arendt CA, Bug G, Serve H, Vogl TJ, Zeiher AM, Carr-White G, Nagel E, Puntmann VO. CMR imaging biosignature of cardiac involvement due to cancer-related treatment by T1 and T2 mapping. Int J Cardiol. 2019 Jan 15;275:179-186. doi: 10.1016/j.ijcard.2018.10.023. Epub 2018 Oct 11. PMID 30360992
- [Derived] de Leuw P, Arendt CT, Haberl AE, Froadinadl D, Kann G, Wolf T, Stephan C, Schuettfort G, Vasquez M, Arcari L, Zhou H, Zainal H, Gawor M, Vidalakis E, Kolentinis M, Albrecht MH, Escher F, Vogl TJ, Zeiher AM, Nagel E, Puntmann VO. Myocardial Fibrosis and Inflammation by CMR Predict Cardiovascular Outcome in People Living With HIV. JACC Cardiovasc Imaging. 2021 Aug;14(8):1548-1557. doi: 10.1016/j.jcmg.2021.01.042. Epub 2021 Apr 14. PMID 33865770